CLINICAL TRIAL: NCT03032289
Title: Association Between Active Transport and Acute Myocardial Infarction: Cross Sectional Ecological Study Using National Registry and Census Data
Brief Title: Association Between Active Transport and Acute Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Marlous Hall, Senior Epidemiologist, University of Leeds
Other Study IDs: UoL_MINAP_Cycling
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Acute Myocardial Infarction
Keywords: active transport; cycling; walking
MeSH Terms: interventions — Biological Transport, Active

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Active Transport — Active transport, most commonly walking or cycling, is the use of physical activity to commute.

SUMMARY:
This study aims to investigate the association between active transport and the incidence of acute myocardial infarction in England.

DETAILED DESCRIPTION:
This is a cross sectional ecological study using aggregated data from the existing Myocardial Ischaemia National Audit Project between 2010 and 2013. Data on active transport according to local authority was obtained from the UK 2001 and 2011 census, whilst important confounders including deprivation levels, prevalence of obesity and population smoking estimates were obtained from Public Health England.

In addition to investigating the association between active transport and AMI, we also studied the extent to which the components of active transport, cycling and walking, were associated with AMI, and investigated whether any associations were contingent on a time lag effect between the dates of exposure to active transport and indecent AMI.

ELIGIBILITY:
Inclusion Criteria:

* All cases of acute myocardial infarction recorded in MINAP between 2003 and 2010

Exclusion Criteria:

* Cases aged <16 and >64 years

Ages: 16 Years to 64 Years | Sex: All
Age Groups: Child, Adult
Study Population: All cases of acute myocardial infarction recorded in the Myocardial Ischaemia National Audit Project (MINAP).
Sampling Method: Non-Probability Sample
Enrollment: 100482 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
Acute myocardial infarction | 2010 to 2013
  Admissions for acute myocardial infarction as recorded in MINAP

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Institute for Data Analytics, Leeds, United Kingdom